CLINICAL TRIAL: NCT00291187
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Study to Investigate the Efficacy and Safety of VEC-162 and Matching Placebo in Healthy Male and Female Subjects With Induced Transient Insomnia
Brief Title: VEC-162 Study in Healthy Adult Volunteers in a Model of Insomnia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VP-VEC-162-3101
Record Dates: First submitted 2006-02-03; First posted 2006-02-13 (Estimated); Results first posted 2014-10-15 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Take orally 30 minutes prior to bedtime.
  Interventions: Drug: Placebo
- 20 mg VEC-162 (Experimental): 20 mg taken orally 30 minutes prior to bedtime.
  Interventions: Drug: 20 mg VEC-162
- 50 mg VEC-162 (Experimental): 50 mg taken orally 30 minutes prior to bedtime.
  Interventions: Drug: 50 mg VEC-162
- 100 mg VEC-162 (Experimental): 100 mg taken orally 30 minutes prior to bedtime.
  Interventions: Drug: 100 mg VEC-162

INTERVENTIONS:
Drug: 20 mg VEC-162 — 20 mg VEC-162
  Arms: 20 mg VEC-162
Drug: 50 mg VEC-162 — 50 mg VEC-162
  Arms: 50 mg VEC-162
Drug: 100 mg VEC-162 — 100 mg VEC-162
  Arms: 100 mg VEC-162
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety and efficacy of VEC-162 compared to placebo to improve sleep parameters in a model of insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects with no medical, psychiatric or current sleep disorders.
* Subject must sign a written consent form.

Exclusion Criteria:

* Recent history of night shift work or jet lag.
* Prior experience sleeping in a sleep lab environment.
* History of sleep disorders.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 411 (Actual)
Dates: Start 2006-02; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vanda Pharmaceuticals, Study Director — Vanda Pharmaceuticals
Locations (19):
- United States (19):
  - Vanda Investigational Site, Birmingham, Alabama
  - Vanda Investigational Site, Phoenix, Arizona
  - Vanda Investigational Site, San Diego, California
  - Vanda Investigational Site, San Francisco, California
  - Vanda Investigational Site, Santa Monica, California
  - Vanda Investigational Site, Miami, Florida
  - Vanda Investigational Site, Naples, Florida
  - Vanda Investigational Site, Pembroke Pines, Florida
  - Vanda Investigational Site, St. Petersburg, Florida
  - Vanda Investigational Site, Atlanta, Georgia
  - Vanda Investigational Site, Overland Park, Kansas
  - Vanda Investigational Site, Chevy Chase, Maryland
  - Vanda Investigational Site, New York, New York
  - Vanda Investigational Site, Rochester, New York
  - Vanda Investigational Site, Raleigh, North Carolina
  - Vanda Investigational Site, Cincinnati, Ohio
  - Vanda Investigational Site, Columbia, South Carolina
  - Vanda Investigational Site, Austin, Texas
  - Vanda Investigational Site, Plano, Texas

REFERENCES:
- [Derived] Rajaratnam SM, Polymeropoulos MH, Fisher DM, Roth T, Scott C, Birznieks G, Klerman EB. Melatonin agonist tasimelteon (VEC-162) for transient insomnia after sleep-time shift: two randomised controlled multicentre trials. Lancet. 2009 Feb 7;373(9662):482-91. doi: 10.1016/S0140-6736(08)61812-7. Epub 2008 Dec 4. PMID 19054552

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place at 20 US sites. The first subject was screened on February 9th 2006, the first subject enrolled on March 10th, 2006, and the last subject completed on August 21st 2006.
Pre-assignment Details: Prior to treatment assignment, subjects were instructed to start a sleep schedule that required staying in bed and trying to sleep for at least 8 hours per night.
  One subject randomized to VEC-162 50 mg was non-compliant for sleep schedule. Subject was discontinued on Day 1 prior to study drug administration.
Groups:
- Placebo: taken orally 30 minutes prior to bedtime
- VEC-162 20 mg: 20 mg taken orally 30 minutes prior to bedtime
- VEC-162 50 mg: 50 mg taken orally 30 minutes prior to bedtime
- VEC-162 100 mg: 100 mg taken orally 30 minutes prior to bedtime
Period: Overall Study
Arm/Group | Placebo | VEC-162 20 mg | VEC-162 50 mg | VEC-162 100 mg
Started | 103 | 100 | 103 | 106
Completed | 103 | 100 | 102 | 106
Not Completed | 0 | 0 | 1 | 0
Not completed — Protocol Violation- No Drug Administered | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-Treat. A total of 411 subjects received treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | VEC-162 20 mg | VEC-162 50 mg | VEC-162 100 mg | Total
Number analyzed (Participants) | 103 | 100 | 102 | 106 | 411
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.9 (7.28) | 30.8 (8.41) | 31.0 (8.51) | 31.2 (8.19) | 31.0 (8.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 62 | 58 | 73 | 261
  Male | 35 | 38 | 44 | 33 | 150

OUTCOME MEASURES:

1. Primary Outcome: Average Improvement of Latency to Persistent Sleep (LPS)
Description: The average improvement in Latency to persistent sleep (the number of minutes between Lights Off and the onset of at least 10 minutes of persistent sleep, as measured by polysomnography) is defined as the difference observed in the VEC-162 treated subjects compared with placebo treated subjects.
Time Frame: Night 1
Population: Modified ITT defined as any subject randomized into the study who received a dose of study drug and had PSG data. For the purposes of this trial, a subject was considered to have PSG data if 50% or more of the full night PSG was scored.
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Placebo | VEC-162 20 mg | VEC-162 50 mg | VEC-162 100 mg
Number analyzed (Participants) | 103 | 100 | 102 | 106
minutes | 45.8 (4.28) | 24.3 (4.35) | 19.6 (4.31) | 23.1 (4.21)
Statistical Analysis 1: Comparison: Placebo vs VEC-162 20 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -21.5, 95% CI 2-sided [-33.1 to -9.9]
Statistical Analysis 2: Comparison: Placebo vs VEC-162 50 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -26.3, 95% CI 2-sided [-37.8 to -14.7]
Statistical Analysis 3: Comparison: Placebo vs VEC-162 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -22.8, 95% CI 2-sided [-34.2 to -11.3]

2. Secondary Outcome: Average Improvement of Wake After Sleep Onset (WASO)
Description: The average improvement of wake after sleep onset (time spent awake between onset of sleep and lights on, determined by PSG) is defined as the difference observed in the VEC-162 treated subjects compared with placebo treated subjects.
Time Frame: Night 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Placebo | VEC-162 20 mg | VEC-162 50 mg | VEC-162 100 mg
Number analyzed (Participants) | 103 | 100 | 102 | 106
minutes | 139.3 (7.33) | 115.1 (7.46) | 105.6 (7.39) | 121.9 (7.22)
Statistical Analysis 1: Comparison: Placebo vs VEC-162 20 mg; Test type: Superiority or Other; p = 0.017, ANCOVA; Mean Difference (Final Values) = -24.2, 95% CI 2-sided [-44.1 to -4.3]
Statistical Analysis 2: Comparison: Placebo vs VEC-162 50 mg; Test type: Superiority or Other; p = 0.001, ANCOVA; Mean Difference (Final Values) = -33.7, 95% CI 2-sided [-53.6 to -13.9]
Statistical Analysis 3: Comparison: Placebo vs VEC-162 100 mg; Test type: Superiority or Other; p = 0.081, ANCOVA; Mean Difference (Final Values) = -17.4, 95% CI 2-sided [-37.0 to 2.1]

3. Post Hoc Outcome: Average Improvement in Total Sleep Time (TST)
Description: The average improvement in Total sleep time (determined by PSG and defined as the number of non-wake minutes between lights off and lights on) is defined as the difference observed in the VEC-162 treated subjects compared with placebo treated subjects.
Time Frame: Night 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Minutes
Arm/Group | Placebo | VEC-162 20 mg | VEC-162 50 mg | VEC-162 100 mg
Number analyzed (Participants) | 103 | 100 | 102 | 106
Minutes | 317.6 (7.65) | 351.4 (7.78) | 365.5 (7.71) | 347.2 (7.53)
Statistical Analysis 1: Comparison: Placebo vs VEC-162 20 mg; Test type: Superiority or Other; p = 0.002, ANCOVA; Mean Difference (Final Values) = 33.7, 95% CI 2-sided [13.0 to 54.5]
Statistical Analysis 2: Comparison: Placebo vs VEC-162 50 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 47.9, 95% CI 2-sided [27.2 to 68.6]
Statistical Analysis 3: Comparison: Placebo vs VEC-162 100 mg; Test type: Superiority or Other; p = 0.005, ANCOVA; Mean Difference (Final Values) = 29.6, 95% CI 2-sided [9.1 to 50.0]

4. Post Hoc Outcome: Average Improvement in Latency to Non-awake (LNA)
Description: The average improvement in latency to non-awake (length of time elapsed between lights off and first epoch of sleep determined by PSG) is defined as the difference observed in the VEC-162 treated subjects compared with placebo treated subjects.
Time Frame: Night 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Minutes
Arm/Group | Placebo | VEC-162 20 mg | VEC-162 50 mg | VEC-162 100 mg
Number analyzed (Participants) | 103 | 100 | 102 | 106
Minutes | 22.3 (2.88) | 11.2 (2.93) | 8.0 (2.90) | 10.0 (2.84)
Statistical Analysis 1: Comparison: Placebo vs VEC-162 20 mg; Test type: Superiority or Other; p = 0.006, ANCOVA; Mean Difference (Final Values) = -11.1, 95% CI 2-sided [-18.9 to -3.3]
Statistical Analysis 2: Comparison: Placebo vs VEC-162 50 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -14.3, 95% CI 2-sided [-22.1 to -6.5]
Statistical Analysis 3: Comparison: Placebo vs VEC-162 100 mg; Test type: Superiority or Other; p = 0.002, ANCOVA; Mean Difference (Final Values) = -12.3, 95% CI 2-sided [-20.0 to -4.6]

ADVERSE EVENTS:
Time Frame: Day 1 through Day 2.
Arm/Group | Placebo | VEC-162 20 mg | VEC-162 50 mg | VEC-162 100 mg
Serious Adverse Events (participants affected / at risk) | 0/103 | 0/100 | 0/102 | 0/106
Other Adverse Events (participants affected / at risk) | 5/103 | 7/100 | 5/102 | 6/106
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=103) | VEC-162 20 mg (N=100) | VEC-162 50 mg (N=102) | VEC-162 100 mg (N=106)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 3 (3) | 3 (3)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Abnormal Dreams (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No